CLINICAL TRIAL: NCT03891680
Title: Comparison Between Intraarticular Botox Injection Versus Genicular Pulsed Radio Frequency in Treatment of Patients With Osteoarthritis
Brief Title: Intra Articular Botox Injection in Treatment of Osteoarthritis
Acronym: Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Botox in osteoarthritis
Record Dates: First submitted 2019-03-23; First posted 2019-03-27 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis Knees Both

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botox injection (Experimental)
  Interventions: Drug: Botox Injectable Product
- Genicular Radio frequency (Active Comparator)
  Interventions: Device: Radiofrequancy

INTERVENTIONS:
Drug: Botox Injectable Product — Intra articular Botox injection
  Arms: Botox injection
Device: Radiofrequancy — Genicular nerves radiofrequancy
  Arms: Genicular Radio frequency

SUMMARY:
Compared the short and long term effects sonography guided of intra articular Botox injection to relief pain and improve patients activity of daily living and disability to genicular nerves pulsed radio frequency fluoroscopy guided

DETAILED DESCRIPTION:
Compared the short and long term effects of sonography guided intra articular Botox injection to relief pain and improve patients activity of daily living and disability to genicular nerves pulsed radio frequency fluoroscopy guided

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis

Exclusion Criteria:

* coagulopathy Organ failure

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Pain visual analog scale | 6 months
  0-10 Visual analog scale( less than 3 no pain 3-5 in pain, more than 5 sever pain

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Allam, Study Chair — Physical medicine Tanta university; Rasha Gaber, Study Chair — Biochemistry Tanta university; Ke Vin, Study Chair — Taiwan
Locations (1):
- Manal Hassanien, Asyut, Egypt